CLINICAL TRIAL: NCT00001117
Title: Dynamics of Hepatitis C Infection in Subjects With Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV) Receiving Highly Active Antiretroviral Therapy (HAART)
Brief Title: A Study to Evaluate the Effects of Anti-HIV Drugs in HIV-Positive Patients Who Also Have Hepatitis C Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 383
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections; Hepatitis C
Keywords: HIV-1; Drug Therapy, Combination; Hepatitis C; RNA, Viral; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Hepatitis C

SUMMARY:
This study evaluates patients infected with both HIV and Hepatitis C virus (HCV) who are receiving anti-HIV drugs. The purpose of this study is to learn more about HCV infection in patients whose HIV blood level decreases to less than 500 copies/ml.

DETAILED DESCRIPTION:
Sixty naive patients with HIV and confirmed hepatitis C who are co-enrolled in another AACTG antiretroviral study that involves the testing of HAART (Highly Active Antiretroviral Therapy) are entered on this prospective study. Patients who are defined as naive have never received specific, active antiretroviral agents that sustain viral suppression below the limit of detection (500 copies/ml) or have received those agents for only a very limited time. HAART is defined as therapy which is likely to result in HIV-1 RNA plasma levels less than 500 copies/ml for at least 16 weeks. Plasma is collected and evaluated during the study for additional quantitative measurements: Hepatitis C virus (HCV) by HCV RNA PCR and HIV-1 RNA levels. All evaluations for HIV-1 RNA are obtained from the co-enrolled study at the following time points: Pre-entry, entry, at least 2 measurements before Week 16, Week 16, and at least 1 measurement after Week 16.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive and have Hepatitis C.
* Have an HIV blood level of at least 2,500 copies/ml 30 days before study entry.
* Are co-enrolled in an active adult AIDS clinical trial using anti-HIV treatment.
* Are at least 13 years of age (parent or guardian consent required if under 18).

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have liver disease.
* Have cancer requiring chemotherapy.
* Have Hepatitis B.
* Abuse alcohol and/or drugs.
* Have received certain antiretroviral (anti-HIV) drugs in the past.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Chung, Study Chair; Cecilia Shikuma, Study Chair
Locations (43):
- United States (42):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Marin County Specialty Clinic, San Rafael, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Chung RT, Evans SR, Yang Y, Theodore D, Valdez H, Clark R, Shikuma C, Nevin T, Sherman KE; AIDS Clinical Trials Group 383 Study Team. Immune recovery is associated with persistent rise in hepatitis C virus RNA, infrequent liver test flares, and is not impaired by hepatitis C virus in co-infected subjects. AIDS. 2002 Sep 27;16(14):1915-23. doi: 10.1097/00002030-200209270-00008. PMID 12351951